CLINICAL TRIAL: NCT04425239
Title: Intermittent or Continuous Panitumumab Plus FOLFIRI for First-line Treatment of Patients With RAS/B-RAF Wild-type Metastatic Colorectal Cancer: a Randomized Phase 2 Trial
Brief Title: Intermittent or Continuous Panitumumab Plus FOLFIRI for RAS/B-RAF Wild-type Metastatic Colorectal Cancer
Acronym: IMPROVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPROVE
Record Dates: First submitted 2020-05-03; First posted 2020-06-11 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer Stage IV
Keywords: metastatic colorectal cancer; RAS and BRAF wild type; intermittent therapy; liquid biopsy; panitumumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTINUOUS ARM: (Active Comparator): Patients will receive Panitumumab plus FOLFIRI until progressive disease, unacceptable toxicity or informed consent withdrawal.
  Interventions: Drug: Panitumumab
- INTERMITTENT ARM: (Experimental): Patients will have a treatment free interval until progressive disease (PD), when they will receive up to 8 cycles of Panitumumab plus FOLFIRI. In the presence of complete or partial response, or stable disease, non-progressing patients will undergo again to treatment free interval until PD, when they will restart treatment. Treatment cycling will continue till any PD on treatment.
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — Continuous administation
  Other Names: Irinotecan; Fluorouracil plus folinic acid
  Arms: INTERMITTENT ARM:
Drug: Panitumumab — Intermittent administation
  Other Names: Irinotecan; Fluorouracil plus folinic acid
  Arms: CONTINUOUS ARM:

SUMMARY:
The investigators hypothesize that intermittent first-line Panitumumab plus FOLFIRI is effective as the same regimen given continuously, in unresectable metastatic RAS and BRAF wild type colorectal cancer patients. Correlative studies on tumor and blood samples could identify potential biomarkers of efficacy and help defining personalized treatment strategy.

DETAILED DESCRIPTION:
This will be a multicenter open label randomized phase II study. The study population will include untreated RAS wild-type metastatic colorectal (mCRC) patients with unresectable disease. A total of 136 patients will be enrolled.

All Patients will receive an induction treatment with panitumumab as 1 hour intravenous infusion at the dosage of 6 mg/kg, given every two weeks, plus FOLFIRI chemotherapy as standard guidelines.

Before start of FOLFIRI plus panitumumab, at the time of enrollment, patients will be immediately randomized electronically 1:1 to one of the two arms. Induction treatment with FOLFIRI plus panitumumab will continue until progressive disease, unacceptable toxicity or informed consent withdrawal, or for up to 8 cycles. At the end of induction treatment, in presence of complete or partial response, or stable disease, non-progressing patients will be allocated to one of the two pre-assigned arms:

A) CONTINOUS: FOLFIRI plus panitumumab until progressive disease, unacceptable toxicity or informed consent withdrawal. Panitumumab will be administered as a 6 mg/kg intravenous infusion over 60 minutes (day 1) every 2 weeks. The dose of Panitumumab should be administered prior to chemotherapy. Irinotecan will be administered as a 180 mg/m2 intravenous infusion over 60 minutes (day 1) every 2 weeks. Folinic acid will be administered as a 200 mg/m2 intravenous infusion over 120 minutes before 5- fluorouracil infusion (day 1) every 2 weeks. 5-fluorouracil will be administered as a 400 mg/m2 intravenous bolus injection (day 1) followed by 2400 mg/m246-hours continuous infusion (day 1), every 2 weeks. Cycle length will be 2 weeks +/- 3 days.

B) INTERMITTENT: treatment free interval until progressive disease; followed by up to 8 cycles of FOLFIRI plus panitumumab; in presence of complete or partial response, or stable disease, non-progressing patients will undergo again to treatment free interval until PD, when they will restart treatment. Treatment cycling will continue till any progressive disease on treatment. Panitumumab will be administered at same dose and infusion with FOLFIRI.

All measurable and non-measurable lesions must be documented at screening (within 21 days prior to randomization) and re-assessed at each subsequent tumor evaluation (every 8 weeks while the patient is on study). Tumor assessment by CT scan of chest, abdomen and pelvis; CEA, CA 19.9; and any other tests having resulted positive during baseline staging, will be performed at week 8 and every 8 weeks thereafter, until disease progression, accordingly with RECIST V 1.1 criteria.

Toxicities will be evaluated throughout the study treatment and graded according to the NCI Common Toxicity Criteria.

The National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTC-AE) Version 4.03 will be used to evaluate the clinical safety of the treatment in this study. Patients will be assessed for AEs at each clinical visit and as necessary throughout the study.

Quality of Life is assessed by the EORTC QLQ-C30, v. 3.0 questionnaire that are completed by patients at baseline, at week 16 and every 8 weeks thereafter.

Biomarkers ancillary study Correlative biological studies will be performed for the evaluation of the biomarkers indicated above on the biological samples available (paraffin-embedded tissue, frozen tissue, blood, serum, etc.). Biomarkers will be evaluated on archival tumor tissues or on newly obtained biopsies at baseline, and during treatment when available. Blood Samples will be collected at baseline, at week 8, 16 and thereafter every 8 weeks concomitantly with tumor assessment.

The sample size is calculated on the basis of median progression-free survival on treatment with intermittent vs continuous Panitumumab plus FOLFIRI, taking into account a median PFS of 11 months observed in the CRYSTAL trial.

The study is designed as a phase II trial with a random assignment to a calibration arm (continous) and to the experimental arm (intermittent). The sample size for intermittent arm is calculated according to the binomial test. The calibration arm has the same sample size, its role is to give a parallel estimation of median PFS to ensure that sample is representative and results are consistent However considering a 5% of drop-outs mainly due to losses to follow-up, the sample size is increased from 130 to 136 patients.

Randomization will be performed with a minimization procedure that will account for center; ECOG (PS 0-1 vs 2); primary site of tumor (Right versus Left); adjuvant treatment (yes vs no); metastatic sites (1 vs>1).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to study procedures and to molecular analyses;
2. Histologically proven diagnosis of colorectal cancer with wildtype RAS and BRAF status in certified laboratories;
3. Initially unresectable metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease;
4. At least one measurable lesion according to RECIST1.1 criteria;
5. Availability of a tumor sample (primary and/or metastatic sites) for exploratory research;
6. Age ≥ 18 years;
7. ECOG PS ≤ 2;
8. Life expectancy of at least 12 weeks;
9. Previous adjuvant chemotherapy allowed only if more than 6 months elapsed between the end of adjuvant and first relapse;
10. Neutrophils ≥ 1.5 x 109/L, Platelets ≥100 x 109/L, Hgb ≥ 9 g/dl;
11. Total bilirubin ≤1.5 time the upper-normal limits (UNL) of the normal values and ASAT (SGOT) and/or ALAT (SGPT) ≤ 2.5 x UNL (or < 5 x UNL in case of liver metastases) alkaline phosphatase ≤ 2.5 x UNL (or < 5 x UNL in case of liver metastases);
12. Creatinine clearance ≥50 mL/min or serum creatinine ≤ 1.5 x UNL;
13. Female with a childbearing potential and male subjects must be willing to use adequate contraception (barrier contraceptive measure, oral contraception, intrauterine device);
14. Will and ability to comply with the protocol.

Exclusion Criteria:

1. Previous treatment for metastatic disease;
2. Radiotherapy to any site within 4 weeks before the study;
3. Any contraindication to use Panitumumab, Irinotecan, 5-FU or folinic acid
4. Known or clinically suspected brain metastases.
5. History or evidence upon physical examination of CNS disease unless adequately treated.
6. Ascites, pleural effusion or pericardial fluid requiring drainage in last 4 weeks.
7. Diagnosis of interstitial pneumonitis or pulmonary fibrosis;
8. Active uncontrolled infections or other clinically relevant concomitant illness contraindicating chemotherapy administration or which, in the investigating physician's opinion, rules out the patient's participation in the study;
9. Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF), serious cardiac arrhythmia requiring medication;
10. Treatment with any investigational drug within 30 days prior to enrolment;
11. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ;
12. Lack of physical integrity of the gastrointestinal tract or history of acute or sub-acute intestinal occlusion or chronic inflammatory bowel disease or chronic diarrhea.
13. Disease that is deemed potentially resectable.
14. Known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs.
15. Any concomitant drugs contraindicated for use with the trial drugs according to the product information of the pharmaceutical companies.
16. Breastfeeding
17. Sexually active males and females (of childbearing potential) unwilling to practice contraception (barrier contraceptive measure or oral contraception) during the study and until 6 months after the last trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2022-04-03 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival | up to 1 year last patients randomized
  Progression Free Survival on treatment (PFSOT) is defined as the time from randomization to the first objective disease progression documented in patients undergoing treatment cycle (objective disease progression during treatment free intervals are excluded) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 1 year last patients randomized
  Overall Survival is defined as the time from randomization to the date of death

OTHER OUTCOMES:
Toxicities | up to 1 year last patients randomized
  Toxicities will be assessed in terms of incidence of Adverse Events (AE) that will be graded according to the NCI CTC-AE Version 4.03 criteria
Assessment of patients'-health-related quality of life | up to 6 months last patients randomized
  Quality of Life will be assessed by the European Organization for Research and Treatment of Cancer [EORTC] QLQ-C30, v.3.0 questionnaire at baseline and at week 12 and 24 during treatment, in both arms
Overall Response Rate | up to 1 year last patients randomized
  Objective Response Rate will be evaluated according to RECIST
Duration of response | up to 1 year last patients randomized
  calculated as the time from the date of the first documented response, complete (CR) or partial (PR), until the date of the first documented progression or death.
Early Tumor Shrinkage | up to 8 weeks last patients randomized
  Early Tumor Shrinkage is defined as the reduction of at least 20% in the sum of longest diameter of the target lesions at week 8 compared with baseline
Depth of response | up to 1 year last patients randomized
  Depth of response is defined as reduction in the sum of longest diameter of the target lesions at the nadir, compared with baseline,in the absence of new lesions or progression of non-target lesions
Genetic Alterations on tumor samples | up to 1 year last patients randomized
  To evaluate the prognostic and predictive value genetic alterations, by next generation sequencing performed on archived tumor samples or on newly obtained biopsies. Analysis is exploratory and will be performed retrospectively after the main study analysis is completed. Analysis will target mainly all relevant clinical mutation in KRAS, NRAS, BRAF, PI3K, EGFR, cKIT and PDGFR genes. Since the identification of new markers correlating with disease activity and the efficacy or safety of treatment are rapidly evolving, the definitive list of analyses remains to be determined; however, it will include a comparative baseline DNA mutational status analysis vs cfDNA
Circulating tumor DNA (liquid biopsy) | up to 1 year last patients randomized
  To evaluate potential biomarkers of primary and secondary resistance analyzing, by Next-generation sequencing, circulating tumor DNA obtained from blood samples ("liquid biopsy") collected at baseline, at week 8, 16 and thereafter every 8 weeks concomitantly with tumor assessment. Analysis of cfDNA mutations on peripheral blood is exploratory and will be performed retrospectively after the main study analysis is completed. Analysis will target mainly all relevant clinical mutation in KRAS, NRAS, BRAF, PI3K, EGFR, cKIT and PDGFR genes. Since the identification of new markers correlating with disease activity and the efficacy or safety of treatment are rapidly evolving, the definitive list of analyses remains to be determined; however, it will include a comparative baseline DNA mutational status analysis vs cfDNA
Metabolomic profiling | up to 1 year last patients randomized
  Metabolomic profiling in peripheral blood at baseline and during treatment evaluated by NMR Spectrometer (600 MHz). The metabolite assignments will be based on the comparison of chemical shifts and spin-spin couplings with reference spectra and tables present in the SBASE-1-1-1 database by AMIX package (Bruker, Biospin, Germany), the human metabolome database (HMDB) and the biological magnetic resonance database (BMRB).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Avallone, MD, Principal Investigator — Istituto Nazionale dei Tumori di Napoli - IRCCS - Fondazione G. Pascale
Locations (1):
- Istituto Nazionale Tumori di Napoli - IRCCS - Fondazione G. Pascale, Napoli, Italy

REFERENCES:
- [Derived] Avallone A, Giuliani F, De Stefano A, Santabarbara G, Nasti G, Montesarchio V, Rosati G, Cassata A, Leo S, Romano C, Tamburini E, Silvestro L, Lotesoriere C, Nappi A, Santini D, Petrillo A, Colombo A, Febbraro A, Leone A, Mannavola F, Laterza MM, Izzo F, Sobrero A, Delrio P, Giannarelli D, Budillon A. Intermittent or Continuous Panitumumab Plus Fluorouracil, Leucovorin, and Irinotecan for First-Line Treatment of RAS and BRAF Wild-Type Metastatic Colorectal Cancer: The IMPROVE Trial. J Clin Oncol. 2025 Mar;43(7):829-839. doi: 10.1200/JCO.24.00979. Epub 2024 Nov 22. PMID 39576946